CLINICAL TRIAL: NCT02794987
Title: Proposal of a Macroscopic Classification for Tissular Lesions of the Bile Duct Detected During Per Oral Cholangioscopy (POCS)
Brief Title: Cholangioscopic Classification of Bile Duct Lesions
Status: Completed | Type: Observational
Sponsor: Instituto Ecuatoriano de Enfermedades Digestivas (Other)
Responsible Party: Sponsor
Other Study IDs: MAY-1-2016
Record Dates: First submitted 2016-05-01; First posted 2016-06-09 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Bile Duct Lesions
Keywords: Bile duct; indeterminate stricture; cholangioscopy; Spyglass

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Histological biopsies of tissular lesions of bile duct
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Classification group: Group of endoscopists that will use the previous classification to select the bile duct tissular lesion images detected by SpyGlass® choledoscopy as benign or malignant with the different subtypes
  Interventions: Device: SpyGlass® choledoscopy
- No classification group: Group of endoscopists that will classified the bile duct tissular lesion images detected by SpyGlass® choledoscopy as benign or malignant with the different subtypes without using the classification.
  Interventions: Device: SpyGlass® choledoscopy

INTERVENTIONS:
Device: SpyGlass® choledoscopy — Stage 1: patients included were evaluated using a standard duodenoscope and both SpyGlass® cholangioscopes: First generation, SpyGlass® Direct Visualization System and Second generation, Digital SpyGlass® DS System (Boston Scientific, Marlborough, Massachusetts, USA) Procedures were performed by one experienced endoscopists with more than 300 ERCP/year (C.R.M). Biopsies were taken in order to correlate to histopathology. Stage 2: patients will be evaluated using a standard duodenoscope and second generation, Digital SpyGlass® DS System (Boston Scientific, Marlborough, Massachusetts, USA). Procedures will be performed by two experienced endoscopists with more than 300 ERCP/year (C.R.M and M.S.A). Biopsies will be taken in order to correlate to histopathology.

SUMMARY:
Endoscopic retrograde cholangio-pancreatography (ERCP) is a diagnostic and therapeutic procedure, however it has an important image limitation. The fluoroscopic cholangiography shows the biliary tree in a two-dimensional view. When an indeterminate biliary stricture is seen, the certainly diagnosis by ERCP depends on a blind biopsy sampling with the risk of missed pathology and sampling errors. SpyGlass® System (Boston Scientific, Marlborough, Massachusetts, USA) is a cholangioscope that enables single-operator, direct visualization of the pancreatico-biliary system and the evaluation of intraductal lesions. It has a digital sensor with 4x resolution and a 1.2 mm working channel that allows the passage of the SpyBite® Forceps biopsy. It has been demonstrated that the use of SpyGlass® System and SpyBite® Forceps changes clinical management in 64% of patients. It has a sensitivity of 76.5% for indeterminate stricture diagnosis, compared to 29.4% and 5.9% sensitivity using blind biopsy brushing catheter respectively. Although it has been described before cholangioscopic images of malignant biliary lesions like an irregular lesion surface with irregular vessels and bleeding or a smooth surface without vessels for benign lesions, there is no current validated classification that allows unify the diagnostic criteria.

Methods: Study design: The study was design to be performed in 2 stages. Stage 1: observational, retrospective study with case collection from September 2013 to September 2015. Patients included had bile duct tissular lesion detected by POCS. The images were correlated to histopathology and 6 month follows up and a classification was finally performed to differentiate benign forma malignant bile duct lesions. Stage 2: patients with bile duct tissular lesion detected by POCS, will be the evaluated in a prospective, non-randomized and double blind manner. Two groups of endoscopist will evaluate the images but only one group will do it using the classification previously performed. Second stage case collection has already started (December 2015) and will include patients until December 2016.

* Endpoint Classification: Efficacy
* Intervention Model: Non interventional
* Primary Purpose: Diagnosis

DETAILED DESCRIPTION:
Setting: Gastroenterology division of the Ecuadorian Institute of Digestive Diseases (IECED), OmniHospital Academic Tertiary Center. The study protocol and consent form has been approved by the Institutional Review Board and will be conducted according to the declaration of Helsinki. Patients will sign an informed consent.

Population selection:

Stage 1: 63 patients enrolled with bile duct tissular lesion detected by POCS. Cholangioscopic lesions images (315) were photographically recorded in order to correlate to, histopathology after targeted or surgical biopsies, and 6 months follow up with POCS. Using the histopathology results, the lesions were classified into benign or malignant. An experienced endoscopist with more than 140 POCS analyzed the images based on the morphological and vascular pattern and performed a POCS macroscopic classification of tissular bile duct lesions as follow: Benign lesions: Type 1 "Villous pattern" (micronodular or villous pattern without vascularity), Type 2 "Polypoid pattern" (adenoma or granuloma pattern without vascularity) and Type 3 "Inflammatory pattern" (regular or irregular fibrous and congestive pattern with regular vascularity). Malignant lesions: Type 1 "Flat pattern" (flat and smooth or irregular surface with irregular or spider vascularity); Type 2 "Polypoid pattern" (polypoid or mass shape with fibrosis and irregular or spider vascularity), Type 3 "Ulcerated pattern" (irregular ulcerated and infiltrative pattern with or without fibrosis and with irregular or spider vascularity) and type 4 "honey-comb pattern" (fibrous honey-comb pattern with or without irregular or spider vascularity).

Stage 2: estimated enrollment of 100 patients with bile duct tissular lesion detected by POCS. Patients included will be analyzed by two groups of endoscopists. One group (classification group) will use the previous classification to select the images as benign or malignant with the different subtypes; and the second group (no classification group or control group) will do it without using the classification.

Endoscopic technique:

Stage 1: patients included were evaluated using a standard duodenoscope (Pentax ED 3670TK, Hoya Co.), the Pentax Video Processor EPK-i5010 and both SpyGlass® cholangioscopes: First generation, SpyGlass® Direct Visualization System and Second generation, Digital SpyGlass® DS System (Boston Scientific, Marlborough, Massachusetts, USA) in a mother-baby manner. Procedures were performed by one experienced endoscopists with more than 300 ERCP/year (C.R.M), in the supine position and under general anesthesia. All patients received antibiotic prophylaxis. Biopsies were taken in order to correlate to histopathology.

Stage 2: patients will be evaluated using a standard duodenoscope (Pentax ED 3670TK, Hoya Co.), the Pentax Video Processor EPK-i7010 and second generation, Digital SpyGlass® DS System (Boston Scientific, Marlborough, Massachusetts, USA) in a mother-baby manner. Procedures will be performed by two experienced endoscopists with more than 300 ERCP/year (C.R.M and M.S.A), in the supine position and under general anesthesia. Half of patients will receive antibiotic prophylaxis because an ongoing cholangioscopic antibiotic prophylaxis protocol. Biopsies will be taken in order to correlate to histopathology.

Inter and intra-observer agreement Stage 1: A data set containing 40 random photographs of the bile duct lesions were presented to 1 expert and 2 non-experts in POCS, whom analyzed the images blindly. Intra and inter-observer reproducibility was measure based on comparison of images between endoscopists.

Stage 2: Intra and inter-observer agreement will be performed in the same manner as stage1.

Statistical analysis: Baseline characteristics will be compared between groups using Chi-square o Fisher Test for categorical variable and Mann-Whitney Test for continuing variables. Accuracy, sensitive, specificity, positive and negative predicts value will be calculated. To examine inter and intra observer agreement, kappa values will be calculated. A P value of less than 0.05 is considered to be statistically significant. All the statistical analysis will be performed using SPSS software suite v.22.

Limitations: the protocol will be performed in only one center.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old patients
* Who agree to participate in the study
* Patients with tissular biliary lesions detected by POCS

Exclusion Criteria:

* Tissular lesions with no histology confirmation (either biopsy or surgical resection in case of malignancy suspicion) or 6 months follow-up by POCS (in case of benign suspicion)
* Severe uncontrolled coagulopathy
* Esophageal, gastric or duodenal stenosing tumors with no possibility of scope passage
* Prior history of esophageal, gastric or surgery with no possibility of scope passage
* Contrast allergy
* Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage 1: 63 patients enrolled with bile duct tissular lesion detected by POCS. Cholangioscopic lesions images (315) were compared to histopathology results and 6 months follow up with POCS, and an experienced endoscopist with more than 140 POCS performed a POCS macroscopic classification of tissular bile duct lesions, based on the morphological and vascular pattern.
  Stage 2: estimated enrollment of 100 patients with bile duct tissular lesion detected by POCS. Patients included will be analyzed by two groups of endoscopists. One group (action group) will use the previous classification to select the images as benign or malignant with the different subtypes; and the second group (control group) will do it without using the classification.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2015-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of vascular and surface features of benign and malignant lesions detected by POCS images, that could be used to perform a macroscopic classification of bile duct tissular lesions | 24 month
  Vascular and surface features were analyzed using POCS images of bile duct lesions and were correlated to histopathology and 6 month follows up. Finally a classification differenciating benign from malignant bile duct lesions, was performed.
The accuracy, sensitivity, specificity, positive and negative predictive value of the macroscopic classification will be measure in order to perform a prospective validation of the classification. | 12 month
  The images of bile duct lesions will be evaluated by two groups of endoscopists but only one will do it using the previously designed classification. Diagnostic accuracy, sensitivity, specificity, positive and negative predictive value will be measure and compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Robles-Medranda, MD, Principal Investigator — Ecuadorian Institute of Digestive Diseases
Locations (1):
- Instituto Ecuatoriano de Enfermedades Digestivas, Omnihospital, Guayaquil, Guayas, Ecuador

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Seelhoff A, Schumacher B, Neuhaus H. Single operator peroral cholangioscopic guided therapy of bile duct stones. J Hepatobiliary Pancreat Sci. 2011 May;18(3):346-9. doi: 10.1007/s00534-010-0360-7. PMID 21480000
- [Background] Tieu AH, Kumbhari V, Jakhete N, Onyimba F, Patel Y, Shin EJ, Li Z. Diagnostic and therapeutic utility of SpyGlass((R)) peroral cholangioscopy in intraductal biliary disease: single-center, retrospective, cohort study. Dig Endosc. 2015 May;27(4):479-485. doi: 10.1111/den.12405. Epub 2014 Dec 11. PMID 25394296
- [Background] Draganov PV, Lin T, Chauhan S, Wagh MS, Hou W, Forsmark CE. Prospective evaluation of the clinical utility of ERCP-guided cholangiopancreatoscopy with a new direct visualization system. Gastrointest Endosc. 2011 May;73(5):971-9. doi: 10.1016/j.gie.2011.01.003. Epub 2011 Mar 17. PMID 21419408
- [Background] Chen YK, Parsi MA, Binmoeller KF, Hawes RH, Pleskow DK, Slivka A, Haluszka O, Petersen BT, Sherman S, Deviere J, Meisner S, Stevens PD, Costamagna G, Ponchon T, Peetermans JA, Neuhaus H. Single-operator cholangioscopy in patients requiring evaluation of bile duct disease or therapy of biliary stones (with videos). Gastrointest Endosc. 2011 Oct;74(4):805-14. doi: 10.1016/j.gie.2011.04.016. Epub 2011 Jul 18. PMID 21762903
- [Background] Draganov PV, Chauhan S, Wagh MS, Gupte AR, Lin T, Hou W, Forsmark CE. Diagnostic accuracy of conventional and cholangioscopy-guided sampling of indeterminate biliary lesions at the time of ERCP: a prospective, long-term follow-up study. Gastrointest Endosc. 2012 Feb;75(2):347-53. doi: 10.1016/j.gie.2011.09.020. PMID 22248602
- [Derived] Robles-Medranda C, Valero M, Soria-Alcivar M, Puga-Tejada M, Oleas R, Ospina-Arboleda J, Alvarado-Escobar H, Baquerizo-Burgos J, Robles-Jara C, Pitanga-Lukashok H. Reliability and accuracy of a novel classification system using peroral cholangioscopy for the diagnosis of bile duct lesions. Endoscopy. 2018 Nov;50(11):1059-1070. doi: 10.1055/a-0607-2534. Epub 2018 Jun 28. PMID 29954008